CLINICAL TRIAL: NCT05141838
Title: Vitamin D Status and Bone Metabolism Status in Children With Congenital Epidermolysis Bullosa
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Medical Research Center for Children's Health, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 307308294
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Bullosa Epidermolysis; Vitamin D Deficiency; Osteoporosis; Osteopenia; Phosphorus and Calcium Disorders
Keywords: Children, Only
MeSH Terms: conditions — Epidermolysis Bullosa; Vitamin D Deficiency; Osteoporosis; Bone Diseases, Metabolic | interventions — Vitamin D; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 - Vitamin D (Experimental): Patients receiving vitamin D supplements in therapy
  Interventions: Drug: Vitamin D
- Group 2 - Oral nutritional supplement (Experimental): Patients receiving oral nutritional supplement
  Interventions: Dietary Supplement: Oral nutritional supplement
- Group 3 - Vitamin D+Oral nutritional supplement (Experimental): Patients receiving vitamin D supplements and oral nutritional supplement in therapy
  Interventions: Drug: Vitamin D; Dietary Supplement: Oral nutritional supplement
- Group 4 - No intervention (No Intervention): Patients with dystrophic form of congenital epidermolysis bullosa who have not taken vitamin D supplements and/or oral nutritional supplement

INTERVENTIONS:
Drug: Vitamin D — Adding vitamin D preparations to the therapy in the individual required dosage to correct the deficient state
  Arms: Group 1 - Vitamin D; Group 3 - Vitamin D+Oral nutritional supplement
Dietary Supplement: Oral nutritional supplement — Adding оral nutritional supplement to the therapy depending on the degree of protein-energy malnutrition
  Arms: Group 2 - Oral nutritional supplement; Group 3 - Vitamin D+Oral nutritional supplement

SUMMARY:
This retrospective prospective study is aimed at studying the level of vitamin D supply and identifying markers of bone tissue remodeling in order to develop approaches to the prevention of osteopenia and osteoporosis in children with congenital epidermolysis bullosa.

DETAILED DESCRIPTION:
This retrospective prospective interventional study will examine vitamin D availability and its relationship with clinical disease, patient gender and age, and season. The mechanisms of impairment of phosphorus-calcium metabolism and bone tissue metabolism will be analyzed on the basis of biochemical parameters and instrumental research methods in children with dystrophic epidermolysis bullosa in order to develop personalized approaches for correcting vitamin D status and bone metabolism disorders in children with epidermolysis bullosa, followed by an assessment of their clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of epidermolysis bullosa;
* Signing by parents (legal representatives) of informed consent to participate in the study and fulfill the requirements of the study

Exclusion Criteria:

* not planned

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2020-11-21 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin D level | Baseline
  Study of the provision of vitamin D in children with dystrophic and simple forms of epidermolysis bullosa based on the level of 25 (OH) vitamin D (25 hydroxycholecalciferol) in the blood
Vitamin D level | 24 week
  Study of the provision of vitamin D in children with dystrophic and simple forms of epidermolysis bullosa based on the level of 25 (OH) vitamin D (25 hydroxycholecalciferol) in the blood
Phosphorus-calcium metabolism assessment | Baseline
  Study of levels of calcium, phosphorus, parathyroid hormone, creatinine, magnesium, albumin in the blood
Phosphorus-calcium metabolism assessment | 24 week
  Study of levels of calcium, phosphorus, parathyroid hormone, creatinine, magnesium, albumin in the blood
Assessment of the state of bone tissue | Baseline
  Study of levels of alkaline phosphatase, osteocalcin, b-CrossLaps, P1NP in the blood
Assessment of the state of bone tissue | 24 week
  Study of levels of alkaline phosphatase, osteocalcin, b-CrossLaps, P1NP in the blood
Assessment of indicators of physical development | Baseline
  Z-score calculation (weight-for-height z-score)
Assessment of indicators of physical development | 24 wee
  Z-score calculation (weight-for-height z-score)

SECONDARY OUTCOMES:
Assessment of bone mineral density | Baseline
  dual-energy X-ray densitometry
Assessment of bone mineral density | 24 week
  dual-energy X-ray densitometry
Bone age assessment | Baseline
  X-ray of the bones of the hand with an assessment of bone age
Bone age assessment | 24 week
  X-ray of the bones of the hand with an assessment of bone age

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Children's Health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided